CLINICAL TRIAL: NCT02478034
Title: Effekte Von Fludrocortison Auf Soziale Kognition Und Gedächtnis Unter Berücksichtigung Von Geschlechtereffekten
Brief Title: Effects of Mineralocorticoid Receptor Stimulation on Cognition
Acronym: MR-STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, Prof. Dr., Head: Clinical Psychology, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WI-CO-2
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Individuality
MeSH Terms: interventions — Fludrocortisone; fludrocortisone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fludrocortisone (Experimental): effects of fludrocortisone on cognition compared to placebo
  Interventions: Other: Fludrocortisone
- Placebo (Placebo Comparator): effects of fludrocortisone on cognition compared to placebo
  Interventions: Other: Fludrocortisone

INTERVENTIONS:
Other: Fludrocortisone — effects of fludrocortisone on cognition compared to placebo
  Other Names: Florinef (Squibb & Sons Limited)

SUMMARY:
In this study the effects of mineralocorticoid stimulation on social cognition will be investigated in healthy young individuals.

DETAILED DESCRIPTION:
80 healthy young individuals (40 females and 40 male) will be recruited an randomized to either placebo or 0.4 mg Fludrocortison before testing. Tasks will on emotion recognition, Task Switch, visual spacial memory and decision making will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* free of medication
* age 18 - 30

Exclusion Criteria:

* any medication
* severe illness

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
social cognition | 25 min
  computer based tests: emotion recognition

SECONDARY OUTCOMES:
memory | 20 min
  computer based test on visuospacial memory
decision making | 25 min
  computer based tests: BART

CONTACTS AND LOCATIONS:
Overall Officials: Katja Wingenfeld, PhD, Principal Investigator — Charité University
Locations (1):
- Charite University, Berlin, Germany